CLINICAL TRIAL: NCT00232583
Title: Preservation of Beta-cell Function in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ildiko Lingvay, MD, MPH, MSCS, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1003-623
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: TYpe 2 diabetes mellitus; Newly diagnosed; Beta-cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Insulin; Pioglitazone; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metfomin and Insulin (Active Comparator): Metformin 1000mg/BID and Insulin Novolog 70/30 per protocol titration
  Interventions: Drug: Metformin; Drug: Insulin
- Metformin, Pioglitazone and Glyburide (Active Comparator): Metformin 1000mg/BID, Pioglitazone 45 mg and glyburide per protocol titration
  Interventions: Drug: Metfomin; Drug: Pioglitazone; Drug: glyburide

INTERVENTIONS:
Drug: Metformin — Metformin 1000mg/BID
  Arms: Metfomin and Insulin
Drug: Insulin — Insulin Novolg 70/30 per protocol titration
  Arms: Metfomin and Insulin
Drug: Metfomin — Metformin 1000mg/BID
  Arms: Metformin, Pioglitazone and Glyburide
Drug: Pioglitazone — Pioglitazone 45mg
  Arms: Metformin, Pioglitazone and Glyburide
Drug: glyburide — Glyburide per protocol titration
  Arms: Metformin, Pioglitazone and Glyburide

SUMMARY:
The study evaluates the rate beta-cell function decline in newly diagnosed type 2 diabetic patients on two different treatment regimens: insulin and metformin versus glyburide, metformin and pioglitazone.

DETAILED DESCRIPTION:
This is a 72 months long randomized clinical trial longitudinally evaluating beta-cell function, as well as glycemic control and inflammatory markers in newly diagnosed type 2 diabetic patients on two different treatment regimens: insulin and metformin versus glyburide, metformin and pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus diagnosed within the prior 2 months
* HbA1c > 7% at the time of inclusion
* willing to perform intensive diabetes management
* able to comply with treatment and follow-up regimen

Exclusion Criteria:

* HbA1c > 8% at time of randomization
* creatinine > 1.5 mg/dl
* liver function tests > 3 times the upper limit of normal
* severe anemia
* severe proliferative retinopathy
* NYHA class III or IV heart failure
* active CAD or recent (within 6 months) MI
* pregnant, willing to get pregnant, or not willing to practice any contraceptive method
* non-english speaking
* active heavy alcohol or illicit drug users (within past 6 months)
* history of lactic acidosis

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Raskin, MD, Principal Investigator — University of Texas; Ildiko Lingvay, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

REFERENCES:
- [Result] Lingvay I, Kaloyanova PF, Adams-Huet B, Salinas K, Raskin P. Insulin as initial therapy in type 2 diabetes: effective, safe, and well accepted. J Investig Med. 2007 Mar;55(2):62-8. doi: 10.2310/6650.2007.06036. PMID 17362692
- [Derived] Harrison LB, Adams-Huet B, Raskin P, Lingvay I. beta-cell function preservation after 3.5 years of intensive diabetes therapy. Diabetes Care. 2012 Jul;35(7):1406-12. doi: 10.2337/dc11-2170. PMID 22723578
- [Derived] Lingvay I, Legendre JL, Kaloyanova PF, Zhang S, Adams-Huet B, Raskin P. Insulin-based versus triple oral therapy for newly diagnosed type 2 diabetes: which is better? Diabetes Care. 2009 Oct;32(10):1789-95. doi: 10.2337/dc09-0653. Epub 2009 Jul 10. PMID 19592630

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at UT Southwestern Clinical Diabetes Research Office
Pre-assignment Details: A 3-months run-in period preceeded randomization. During this period all patients were treated with insulin and metformin.
Groups:
- Metfomin & Insulin: Insulin NovoLog 70/30 BID adjusted to target fasting blood glucose level of 70 to 110 mg/dL and postprandial blood sugar < 140 mg/dL and Metformin 2,000 mg/day (or maximum tolerated dose).
- Metfomin, Pioglitazone & Glyburide: Metformin 2,000 mg (or maximum tolerated dose); glyburide 1.25 mg BID and 15 mg daily pioglitazone (pioglitazone was titrated monthly to a final dose of 45 mg daily).
Period: Overall Study
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Started | 29 | 29
Completed | 19 | 16
Not Completed | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (9.7) | 45.0 (10.7) | 44.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 20 | 17 | 37
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Beta-cell Function - C-peptide AUC (Area Under the Curve)
Description: C-peptide AUC during a 3-hours mixed meal challenge testing
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: ng*min/mL
Groups:
- Metformin & Insulin: Insulin NovoLog 70/30 BID adjusted to target fasting blood glucose level of 70 to 110 mg/dL and postprandial blood sugar < 140 mg/dL and Metformin 2,000 mg/day (or maximum tolerated dose).
- Metformin, GLyburide & Pioglitazone: Metformin 2,000 mg (or maximum tolerated dose); glyburide 1.25 mg BID and 15 mg daily pioglitazone (pioglitazone was titrated monthly to a final dose of 45 mg daily).
Arm/Group | Metformin & Insulin | Metformin, GLyburide & Pioglitazone
Number analyzed (Participants) | 29 | 29
ng*min/mL | 2096 (795) | 1725 (618)

2. Secondary Outcome: Insulin Sensitivity as Measure be Matsuda Index
Description: C-peptide-based Matsuda index using following formula: Matsuda index = 500,00 / root square [(fasting c-peptide x fasting glucose x 333) x (average c-peptide 0-120 mins x average glucose 0-120 mins x 333). Higher the Matsuda index, better the insulin sensitivity.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
index | 3.12 (2.62) | 2.45 (1.09)

3. Secondary Outcome: Bet-cell Function Measured by Disposition Index
Description: Disposition index was measured by multiplying the insulin secretion (C-peptide AUC/C-peptide AUC glucose) by the Matsuda index. Disposition index reflects the beta-cell function adjusted for total body insulin sensitivity
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
index | 0.12 (0.07) | 0.16 (0.09)

4. Secondary Outcome: Weight
Description: Body Weight
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Metfomin and Insulin: Insulin NovoLog 70/30 BID adjusted to target fasting blood glucose level of 70 to 110 mg/dL and postprandial blood sugar < 140 mg/dL and Metformin 2,000 mg/day (or maximum tolerated dose).
- Metformin, Pioglitazone and Glyburide: Metformin 2,000 mg (or maximum tolerated dose); glyburide 1.25 mg BID and 15 mg daily pioglitazone (pioglitazone was titrated monthly to a final dose of 45 mg daily).
Arm/Group | Metfomin and Insulin | Metformin, Pioglitazone and Glyburide
Number analyzed (Participants) | 29 | 29
kg | 107.7 (31.1) | 107.9 (31.4)

5. Secondary Outcome: Inflammatory Markers - hsCRP
Description: Inflammatory markers - hsCRP (C reactive protein)
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
mg/L | 6.9 (7.7) | 6.1 (8.9)

6. Secondary Outcome: Inflammatory Markers -Fibrinogen
Description: Inflammatory markers - Fibrinogen
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
mg/dL | 399.0 (82.6) | 395.4 (98.5)

7. Secondary Outcome: Inflammatory Markers - PAI-1
Description: Inflammatory markers - PAI-1 (Plasminogen activator inhibitor type 1)
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
IU/L | 13.9 (11.7) | 16.7 (18.0)

8. Secondary Outcome: Quality of Life Survey (QoL) - Current Health Perception
Description: Current health perception was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 = much better than 3 months ago; 2 - Somewhat better now than 3 months ago; 3 - About the same; 4 - Somewhat worse now than 3 months ago; 5 Much worse now than 3 months ago.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a scale | 2.7 (0.9) | 2.9 (0.9)

9. Secondary Outcome: Quality of Life Survey (QoL) - Treatment Satisfaction
Description: Treatment satisfaction was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 - very satisfied; 2 - moderately satisfied; 3 - neither satisfied nor dissatisfied; 4 - moderately dissatisfied; 5 - very dissatisfied.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a scale | 1.7 (0.5) | 2.1 (0.8)

10. Secondary Outcome: Quality of Life Survey (QoL) - Treatment Impact
Description: Treatment impact was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 - very satisfied; 2 - moderately satisfied; 3 - neither satisfied nor dissatisfied; 4 - moderately dissatisfied; 5 - very dissatisfied.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a sale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a sale | 1.7 (0.2) | 1.8 (0.3)

11. Secondary Outcome: Quality of Life Survey (QoL) - Social or Vocational Worry
Description: Social or vocational worry was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 0-5, where 0 - does not apply; 1 - never; 2 - seldom; 3 - sometimes; 4 - often; 5 - all of the time.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a scale | 1.8 (0.3) | 1.7 (0.3)

12. Secondary Outcome: Quality of Life Survey (QoL) - Hypoglycemia Fear
Description: Hypoglycemia fear was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1-5, where 1 - never worry; 2 - rarely water; 3 - sometimes worry; 4 - often worry; 5 - very often worry
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a scale | 1.8 (0.3) | 1.8 (0.4)

13. Secondary Outcome: Quality of Life Survey (QoL) - Glycemia Control Perception
Description: Glycemia control perception was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a scale score of 1-7, where 1 - extremely controlled and 7 - not at all controlled.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a scale | 2.8 (2.8) | 2.0 (2.0)

14. Secondary Outcome: Quality of Life Survey (QoL) - Lifestyle Flexibility
Description: Lifestyle flexibility was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1 to 5, where 1 - a great deal of choice; 2 - a lot of choice; 3 - some choice; 4 - a little choice; 5 - no choice.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a scale | 2.1 (0.6) | 2.0 (0.6)

15. Secondary Outcome: Quality of Life Survey (QoL) - Social Stigma
Description: Social stigma was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a Likert scale score of 1 to 5, where 1- strongly agree; 2 - somewhat agree; 3 - neither agree nor disagree; 4 - somewhat disagree; 5 - strongly disagree.
Time Frame: 72 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Number analyzed (Participants) | 29 | 29
score on a scale | 2.2 (1.2) | 2.2 (1.7)

16. Secondary Outcome: Quality of Life Survey (QoL) - Satisfaction With Insulin Treatment
Description: Satisfaction with insulin treatment was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a scale score of 1 to 7, where 1 extremely satisfied to 7 - not at all satisfied.
Time Frame: 72 months
Population: Data were not collected from participants in the "Metfomin, Pioglitazone & Glyburide" Arm/Group since patients did not receive insulin.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin
Number analyzed (Participants) | 29
score on a scale | 1.2 (0.9)

17. Secondary Outcome: Quality of Life Survey (QoL) - Willingness to Continue Insulin Treatment
Description: Willingness to continue insulin treatment was measured at randomization and 72 months later using the modified Diabetes Quality of Life Clinical Trial Questionnaire. This questionnaire addresses several areas with respect to diabetes QoL. Answers are in the form of a scale score of 1 to 7, where 1 extremely willing to 7 - not at all willing.
Time Frame: 72 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metfomin & Insulin
Number analyzed (Participants) | 29
score on a scale | 1.4 (0.7)

ADVERSE EVENTS:
Arm/Group | Metfomin & Insulin | Metfomin, Pioglitazone & Glyburide
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/29
Other Adverse Events (participants affected / at risk) | 5/29 | 6/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metfomin & Insulin (N=29) | Metfomin, Pioglitazone & Glyburide (N=29)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) — Cardiac arrest leading to sudden death.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metfomin & Insulin (N=29) | Metfomin, Pioglitazone & Glyburide (N=29)
GI disturbance (Gastrointestinal disorders) | 5 (15) | 6 (18) — Gastrointestinal adverse events included the following conditions: nausea, diarrhea, flatulence and or vomiting. These events were not reported separately.

LIMITATIONS AND CAVEATS:
Relatively small trial, but longest (6-year) follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No